CLINICAL TRIAL: NCT00371605
Title: An Assessment of Voriconazole Pharmacokinetics and Pharmacogenetics in Liver Transplant Recipients - Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Enrolled requested number of patients and completed study. In analysis
Sponsor: University of Pittsburgh (Other)
Other Study IDs: IRB# 0607030
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Liver Transplant; Fungal Infection
Keywords: Voriconazole; Liver Transplant; Fungal Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.

SUMMARY:
A fixed-dosing regimen of voriconazole is routinely used as prophylaxis against aspergillosis in liver transplant patients admitted to the transplant intensive care unit at UPMC. We hypothesize that use of a fixed-dosing regimen of voriconazole will lead to a large degree of variability in drug exposure among liver transplant patients due to: 1) variability in absorption and elimination caused by physiological characteristics unique to this patient population 2) its non-linear pharmacokinetics and 3) the potential for polymorphism in the genes that encode for cytochrome P-450 enzymes that metabolize voriconazole. This is a pilot clinical pharmacokinetic evaluation that will: 1) characterize the plasma concentration versus time profile of voriconazole in liver transplant patients receiving a fixed-dosing regimen to assess for extremes in systemic exposure 2) determine the oral bioavailability of voriconazole in liver transplant patients 3) assess for functionally significant allelic variation of the cytochrome P-450 enzymes that metabolize voriconazole (CYP2C9, CYP2C19 and CYP3A4/5) in both recipient blood and allograft tissue that may contribute extremes in systemic exposure among liver transplant patients. This evaluation will allow for an assessment of the adequacy of the prophylactic regimen in achieving therapeutic drug concentrations in all subjects. Additionally, the utility of genotyping as a clinical tool to identify patients at risk for extremes in voriconazole exposure will be evaluated. The characterization of the pharmacokinetics in liver transplant patients may be utilized to define an optimal therapeutic regimen that will be individualized to target specific concentrations to maximize efficacy and minimize side-effects.

DETAILED DESCRIPTION:
All liver transplant patients receiving voriconazole prophylaxis are eligible to participate in this study. We propose a single-center, observational study in 15 liver transplant patients who are admitted to the ICU and receiving voriconazole prophylaxis as part of standard care. Each patient will undergo blood sampling (27 mL) on one occasion (Pharmacokinetic Study I), while receiving oral voriconazole. A small portion of blood (1 mL) collected during this blood sampling period will be retained for genotyping (specific aim III).

Voriconazole prophylaxis is most often administered to liver transplant patients via the oral route (200 mg twice daily). However, circumstances may arise necessitating the administration of intravenous doses of voriconazole for a subset of patients, as part of their standard care. . Thus, these patients will undergo blood sampling on a maximum two additional occasions: 1) surrounding an intravenous dose dose (27 mL) 2) surrounding an oral dose (27 mL) .

The amount of voriconazole present in the blood samples will be measured via high pressure liquid chromatography. Individual plasma concentration time profiles will be determined following oral and intravenous dosing, respectively. Pharmacokinetic parameter estimates will be derived via population and individual pharmacokinetic data analysis.

The use, dose, and frequency of the medication voriconazole is up to the clinical staff. We will not be altering the delivery, dose or use of the drug. Therefore we cannot provide you with the requested information because it will all depend on the clinical team. We are not intervening to enroll subjects. Subjects will only be enrolled if they are placed on voriconazole and they agreed to participate.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive male or female liver transplant recipients, 18 years old, who are initiated on the voriconazole prophylactic regimen by their transplant physician as part of their standard care, will be eligible for inclusion in the study.

Exclusion Criteria:

* Transplant recipients receiving voriconazole to treat an active fungal infection will be excluded. Transplant recipients that are concurrently receiving medications that are documented to affect voriconazole pharmacokinetics will be excluded. The agents included, but may not be limited to the following; carbamazepine, phenytoin, omeprazole, rifabutin, rifampin, ketoconazole, itraconazole, fluconazole, St. John's wort extract. Those who require therapy with protease inhibitors for human immunodeficiency virus (HIV) infection may be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver transplant patients getting voriconazole clinically
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2006-12; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blair Capitano, Pharm D, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States